CLINICAL TRIAL: NCT02672527
Title: A Randomized Phase III Trial Comparing Trabectedin (Yondelis®) to the Best Supportive Care in Patients With Advanced Soft Tissue Sarcoma
Brief Title: Trial Comparing Trabectedin to the Best Supportive Care in Patients With Sarcoma
Acronym: TSAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-003176-23; 2014/2154 (Other: CSET number)
Record Dates: First submitted 2015-05-06; First posted 2016-02-03 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRA (Experimental): At Day 1 (D1), premedication with dexamethasone (20 mg) and a 5-HT3 receptor antagonist anti-emetic agent will be intravenously administered 30 minutes prior to trabectedin administration. Trabectedin will be administered through a central venous catheter at a starting dose of 1.5 mg/m² over 24 hours, diluted in at least 500 mL of normal saline solution or of glucose 5% injectable solution.
  Each treatment cycle will last 21 days. Treatment duration: the treatment might be pursued until disease progression according to RECIST 1.1, or patient refusal, or toxicities.
  In case of disease progression, the further treatments will be based on investigator's judgement.
  Interventions: Drug: Trabectedin; Drug: Dexamethasone
- BSC (No Intervention): Treatment:
  Patients will receive the best supportive care (BSC) in order to alleviate their symptoms and improve their Quality of Life (QoL).
  Antineoplastic agents (including surgery, radiotherapy, thermotherapy, chemotherapy, immunotherapy, hormonal treatment or antibodies-based treatments) are prohibited.
  Treatment duration: the treatment might be pursued until disease progression according to RECIST 1.1, or patient refusal.
  In case of disease progression, a treatment with trabectedin will be proposed (cross-over). In case of patient refusal, the further treatments will be based on investigator's judgement.

INTERVENTIONS:
Drug: Trabectedin
  Other Names: Yondelis
  Arms: TRA
Drug: Dexamethasone
  Arms: TRA

SUMMARY:
As the transparency committee of the Haute Autorité de Santé pointed out due to lack of data regarding comparative trial of Yondelis versus best supportive care, activity of Yondelis in soft tissue sarcoma remain to be assessed.

For an antineoplastic drug toxicity is moderate. As previous studies shown, overall survival data for patients with advanced or metastatic STS are of poor prognosis despite improvement of results this last years. For example, median overall survival increased from 12,3 months (1987-1991) to 11,4 months (1992-1996) and then 18 months (2002-2006).

Considering the latest results with and without Trabectedin, the investigators may consider that comparing Trabectedin with best supportive care is ethically acceptable as long as patients consent to enter the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood, agreed and signed
2. Tolerance of the central venous line that will be used for Trabectedin infusions.
3. Pathologically confirmed diagnosis of STS at the investigator centre level (and confirmed by Rrepps Network), except the following cases :

   * Low grade fibromyxoid sarcoma (LGFMS),
   * Giant Cells Fibroblastoma,
   * Dermatofibrosarcoma protuberances (DFSP),
   * Angiomatoid fibrous histiocytoma,
   * Alveolar Rhabdomyosarcoma and Embryonal Rhabdomyosarcoma,
   * Mesenchymal and Non-Mesenchymal Chondrosarcoma,
   * Extraskeletal Ewing Sarcoma / Primitive Neuroectodermal Tumour (PNET),
   * Desmoplastic small round-cell tumour (DSRCT ),
   * Gastro-Intestinal Stromal Tumour (GIST),
   * Endometrial Stroma Sarcoma,
   * Osteosarcoma.
4. Histological samples available for centralised histopathological diagnosis and the appropriate genetic diagnosis.
5. Patient who already received no more than 3 previous therapy lines. Therefore, trabectedin might be administered as a 2nd, 3rd or 4th therapy line in case of metastatic STS.
6. Measurable disease as per RECIST (Response Evaluation Criteria In Solid Tumors), and confirmed based on objective data within 14 days prior to study inclusion.
7. Disease progression according to RECIST 1.1 confirmed by imaging evaluation within 14 days prior to study inclusion comparatively to imaging within the previous 6 months.
8. ECOG (Eastern Cooperative Oncology Group) Performance score: 0 or 1.
9. Normal cardiac function as assessed by cardiac ultrasound examination or by MUltiple Gated Acquisition scan (MUGA scan).
10. Biological laboratory parameters meeting the following criteria within 14 days prior to study inclusion:

    * neutrophil leucocytes ≥ 1500 /μL,
    * haemoglobin ≥ 9,0 g/100 mL,
    * platelet count 100 x 103 /μL
    * AST (aspartate aminotransferase) ≤ 2.5 times the investigator local laboratory upper normal limit (UNL),
    * ALT (alanine aminotransferase) ≤ 2.5 times the investigator local laboratory UNL,
    * Alkaline phosphatases ≤ 2.5 UNL,
    * bilirubin ≤ UNL ,
    * CPK ≤ 2.5 times the investigator laboratory UNL,
    * albumin ≥ 25 g/L
    * creatinine clearance measured or calculated (Cockcroft-Gault formula) ≥ 30 mL/min.
11. Patient having reached the majority age at the time they sign the informed consent.
12. Life expectancy of at least 3 months at study entry.
13. Patient covered by the health insurance system.
14. All women of childbearing potential must have a negative serum pregnancy test within 14 days prior to study inclusion.

Exclusion Criteria:

1. Hypersensitivity, history of allergic reaction to trabectedin
2. History of allergic reaction or known hypersensitivity to dexamethasone or to anti-emetic agents belonging to the triptan family (i.e., 5-HT3 receptor antagonists).
3. History of allergic reaction or known hypersensitivity to contrast agents (except if the patient's tumour can be evaluated using MRI without contrast agents).
4. Severe concomitant disease (such as pulmonary fibrosis, interstitial pneumonitis, renal insufficiency, liver failure, cerebrovascular disease, malignant disease requiring blood transfusions, or uncontrolled diabetes).
5. Clinically significant abnormalities of the electrocardiogram test, or one of the following clinically significant cardiac diseases :

   * Congestive cardiac insufficiency,
   * Active coronary disease,
   * Arrhythmia poorly controlled by medicinal products only,
   * Myocardial infarction within one year prior to study entry.
6. Surgery under general anaesthesia within 28 days prior to study entry, exploratory surgery (thoracotomy or laparotomy) within 28 days prior to study entry,.
7. Treatment with one of the following anticancer agents prior to study entry :

   * hormonotherapy within 14 days prior to study entry,
   * other anticancer treatment (such as chemotherapy, targeted therapy, or biological advanced therapy) within 21 days prior to study entry.
8. Radiotherapy within 21 days prior to study entry.
9. History of graft transplantation or stem cell transplantation.
10. Adverse reaction to a previous treatment, other than alopecia, long-lasting, and of grade ≥ 2 severity according to CTCAE (v. 4.0) criteria.
11. Intercurrent infection requiring a systemic antimicrobial treatment (e.g., associated with fever ≥ 38° C),
12. Patients HIV positive and/or viral anti-therapy and/or hepatitis B and/or C. Systematic serology to check the status is not necessary.
13. Brain metastasis, either symptomatic or requiring a treatment.
14. History of another cancer within 5 years prior to study entry (except intra-epithelial neoplasm or basocellular cancer, if they are cured, e.g., thanks to surgical resection or radiotherapy).
15. Psychiatric disorders disturbing the informed consent process.
16. Pregnant or breast-feeding woman; man or woman not complying to contraceptive measures during the following time periods:

    * For the men, during the full study up to 5 months after the last study treatment administration;
    * For the women, femmes, during the full study up to 3 months after the last study treatment administration.
17. Other investigational treatment within 28 days prior to study entry.
18. Prior treatment with trabectedin.
19. Any clinical conditions not compatible with an adequate study conduct, according to investigator's judgement.
20. Patient under administrative or legal supervision, patient hospitalised without his/her consent or for other purposes than research, patient under guardianship or curators, or unable to express his/her consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Assessed every three weeks after randomization then every six weeks until progression or death of any cause whichever came first up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France